CLINICAL TRIAL: NCT01060930
Title: Diesel Exhaust Inhalation, Systemic Nitric Oxide Inhibition and Cardiac Output
Acronym: DISCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DISCO
Record Dates: First submitted 2010-01-28; First posted 2010-02-02 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-04

CONDITIONS: Vascular Function in Healthy Volunteers
Keywords: Nitric oxide; Diesel exhaust; Air pollution; Cardiac output; Healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diesel exhaust exposure (Experimental): 1 hour exposure to dilute diesel exhaust ~ 300 mcg/m3 - during intermittent exercise
  Interventions: Drug: Intravenous infusion of L-NMMA and Nor-epinephrine
- Air exposure (Experimental): 1 hour exposure to filtered air during intermittent exercise
  Interventions: Drug: Intravenous infusion of L-NMMA and Nor-epinephrine

INTERVENTIONS:
Drug: Intravenous infusion of L-NMMA and Nor-epinephrine — Intravenous infusion of 3mg/kg L-NMMA (L-NG-monomethyl arginine; NO synthase inhibitor) and nor-epinephrine at 50 ng/kg/min. Each infusion to run over 15 mins and separated by 45 min to allow return to baseline. Drugs infused in a randomised order. During the study, blood pressure will be measured invasively using an intra-arterial radial artery cannula, central arterial stiffness measured using peripheral arterial tonometry and cardiac output using thoracic bioimpedance.
  Other Names: L-NMMA: Clinalfa Basic, Bachem, Germany

SUMMARY:
Exposure to combustion-derived fine particulate air pollution is associated with cardiovascular mortality and morbidity. In previous studies, exposure to diesel exhaust (a major constituent of urban particulate air pollution) has been shown to impair two important functions of the vascular endothelium: vascular vasomotor function and endogenous fibrinolysis. Our subsequent studies suggest this impairment of vascular function is mediated by a reduction in nitric oxide bioavailability. In this study we aim to investigate the cardiovascular responses to systemic nitric oxide synthase inhibition following exposure to dilute diesel exhaust.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Non smokers
* No regular medication (except oral contraceptive)
* No recent respiratory tract infection (within 6 weeks)

Exclusion Criteria:

* History of asthma or respiratory disease
* Smoking history
* Pregnancy (positive urinary pregnancy test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Blood pressure response to NO inhibition | Blood pressure will be measured continuously through the vascular study using intra-arterial monitoring

SECONDARY OUTCOMES:
Heart rate response to systemic nitric oxide inhibition | Heart rate will be measured continuously throughout the study period using continous electrocardiography
Central arterial stiffness following NO inhibition | Measured at baseline, and every 5 minutes during the 2-hour vascular study
Cardiac output during NO inhibition | Measured at baseline, and every 5 minutes during the 2-hour vascular study
Plasma nitrite (NO) concentrations | Measured at baseline, and every 15 minutes during the 2-hour vascular study
Platelet activation and platelet-monocyte binding | Measured at baseline, and every 30 minutes during the 2-hour vascular study
Heart rate variability | Heart rate will be measured continuously throughout the study period using continous electrocardiography, and HRV subsequently determined for the whole study period and the 2-hour vascular study separately

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy P Langrish, MB BCh MRCP, Principal Investigator — University of Edinburgh
Locations (1):
- University Hospital Umeå, Umeå, Sweden

REFERENCES:
- [Derived] Langrish JP, Unosson J, Bosson J, Barath S, Muala A, Blackwell S, Soderberg S, Pourazar J, Megson IL, Treweeke A, Sandstrom T, Newby DE, Blomberg A, Mills NL. Altered nitric oxide bioavailability contributes to diesel exhaust inhalation-induced cardiovascular dysfunction in man. J Am Heart Assoc. 2013 Feb 19;2(1):e004309. doi: 10.1161/JAHA.112.004309. PMID 23525434